CLINICAL TRIAL: NCT03359005
Title: Irinotecan and Temozolomide for Advanced Ewing Sarcoma After Failure of Standard Multimodal Therapy
Brief Title: Irinotecan and Temozolomide for Ewing Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-EWS-01
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Ewing Sarcoma
Keywords: Ewing Sarcoma; Irinotecan; Temozolomide
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Vincristine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5d VIT (irinotecan, temozolomide and vincristine) (Experimental): Irinotecan 50mg/m2/d IV over 60 minutes on days 1-5.
  Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Vincristine; Drug: Temozolomide
- 5d x 2 VIT (irinotecan, temozolomide and vincristine) (Active Comparator): Irinotecan 20mg/m2/d IV over 60 minutes on days 1-5 and 8-12.
  Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Vincristine; Drug: Temozolomide

INTERVENTIONS:
Drug: Vincristine — vincristine 1.5mg/m2 iv D1,D8
  Other Names: VCR
Drug: Temozolomide — Temozolomide 100mg/m2/d iv on days 1-5.
  Other Names: Temodar

SUMMARY:
The investigators explored the activity of vincristine and irinotecan combined with temozolomide (VIT) in patients with relapsed and metastatic Ewing Sarcoma.

DETAILED DESCRIPTION:
After standard multimodal therapy, the prognosis of relapsed and metastatic Ewing Sarcoma is dismal and unchanged over the last decades. The anti-tumor activity of VIT was demonstrated by several studies in the past. However, the detailed schedule of VIT was not decided. Thus, the investigators explored the activity of 5-d shorter schedule of VIT and 5-d x2w longer schedule of VIT in patients with relapsed and metastatic Ewing Sarcoma after the failure of first-line chemotherapy with doxorubicin, vincristine, cyclophosphamide, ifosphamide and etoposide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Ewing sarcoma.
* Evidence of Ewing sarcoma translocation by fluorescence in situ hybridization (FISH) or real-time polymerase chain reaction (RT-PCT).
* Recurrent or refractory tumors with no known curative treatment options according to the judgment of the investigator.
* Prior treatment consisted of standard Ewing Sarcoma chemotherapy agents including doxorubicin, vincristine, cyclophosphamide, ifosfamide and etoposide; metastatic relapsed and unresectable progressive disease (PD);
* Life expectancy of ≥ 3 months.
* Eastern Cooperative Oncology Group performance status 0-1
* Measurable disease on CT or MRI by RECIST 1.1.
* Adequate organ function.
* Time elapsed from previous therapy must be ≥ 3 weeks for systemic therapy, ≥ 2 weeks for radiation therapy or major surgery.
* Patients who have undergone autologous hematopoietic stem cell transplantation are eligible once they have recovered from all toxicities from therapy.
* Patients who have received allogeneic hematopoietic stem cell transplantation will be eligible 6 months after the procedure provided there is no evidence of active graft-versus-host disease and immunosuppressive treatment has been discontinued for at least 30 days.
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of central nervous system metastatic disease, have been off glucocorticoids for at least 4 weeks, have no overt evidence of neurological deficit and are ≥ 6 weeks from completion of brain irradiation.
* Females of childbearing potential as well as males and their partners must agree to use an effective form of contraception during the study and for 6 months following the last dose of study medication.

Exclusion Criteria:

* Clinically significant unrelated illness which would, in the judgment of the treating physician, compromise the patient's ability to tolerate the investigational agent or be likely to interfere with the study procedures or results.
* Patients with baseline corrected QT interval(QTc) > 480 msec.
* Known hypersensitivity to any of the components of niraparib or prior hypersensitivity reactions to that class of drugs.
* Known hypersensitivity reaction to temozolomide or any of its components, or dacarbazine (DTIC) or any of its components, and irinotecan or any of its components.
* Concomitant use of any other investigational or anticancer agent(s).
* Pregnant patients or patients who are breast feeding. Subjects capable of pregnancy (post menarche and not post-menopausal, defined as over 12 months since final menstrual period) must have a negative pregnancy test within 7 days prior to first dose.
* Inability to swallow capsules.
* Other clinically significant malignant disease diagnosed within the previous 5 years, excluding intra-epithelial cervical neoplasia or non-melanoma skin cancer.
* Known persistent (> 4 weeks) ≥ Grade 2 neutropenia, ≥ Grade 2 thrombocytopenia or > Grade 3 anemia from prior cancer therapy.
* Other kinds of malignant tumors at the same time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2022-11-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Object response rate(ORR) at 12 weeks | 4 months
  complete response (CR) + partial response (PR) at 12 weeks

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  Calculated from the date of treatment start until the time of disease progression or death, whichever comes first.
Overall survival(OS) | 2 years
  Calculated from the date of treatment start until last follow-up or death, whichever comes first.
Duration of response(DOR) | 2 years
  Duration of response is calculated from the day of first response assessment until either progression/death (event) or last day of follow-up (censored).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Ph.D, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided